CLINICAL TRIAL: NCT03283800
Title: Impact of Copper Compression Stockings on Venous Insufficiency and Lipodermatosclerosis: a Randomised Controlled Trial
Brief Title: Copper Impact on Venous Insufficiency and Lipodermatosclerosis
Acronym: CIVIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croydon Health Services NHS Trust (Other)
Responsible Party: Principal Investigator, Mr Abdul H Sultan, Consultant Obstetrician and Gynaecologist, Croydon Health Services NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15/04
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Lipodermatosclerosis; Chronic Venous Insufficiency; Venous Insufficiency; Varicose Veins
Keywords: Copper Oxide; Compression Therapy; Chronic Venous Disease; Randomised Controlled Trial; Lipodermatosclerosis
MeSH Terms: conditions — Lipodermatosclerosis; Venous Insufficiency; Varicose Veins

STUDY DESIGN:
Intervention Model Description: All participants will be asked to wear compression stockings. One of the pair will have copper oxide ions permanently attached to the nylon fibres and these stockings will contain 2-3% copper ions. The participants will wear a copper stocking on one leg (study leg) and a non-copper stocking on the other (control leg).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All stockings are marked with an 'L' for the left or 'R' for the right foot. The manufacturer has randomly marked the copper stockings with an 'L' or 'R' and paired these with a non-copper stocking. A closed envelope will contain the unique numbers of all the pairs of stockings and the information on which stocking contains the copper. This envelope will remain closed for the whole recruitment period and throughout analysis of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copper impregnated compression stocking (Experimental): Copper compression stocking containing 2-3% copper ions to be worn on one leg, daily for 8 weeks.
  Interventions: Other: Copper impregnated compression stocking
- Normal compression stocking (Placebo Comparator): Similar compression stocking without copper to be worn on the other leg, daily for 8 weeks
  Interventions: Other: Normal compression stocking

INTERVENTIONS:
Other: Copper impregnated compression stocking — Copper impregnated compression stocking
  Arms: Copper impregnated compression stocking
Other: Normal compression stocking — Normal compression stocking without copper
  Arms: Normal compression stocking

SUMMARY:
Venous disease has an adverse impact on the quality of life of patients and the NHS spends considerable resources on this chronic condition. Copper has been shown to promote new blood vessel formation and therefore improve blood supply to the affected area and possibly skin conditions. Copper has also been shown to have strong antimicrobial properties. We plan to perform a study whereby patients who would normally be given leg stockings will be asked to wear similar stockings except that one of the stockings will contain copper fibers. Neither the patient nor the clinician will know which is which. Photographs of the leg conditions will be taken at baseline, 2, 4 and 8 weeks to evaluate healing. Benefit will be evaluated by a symptom questionnaire, severity scoring tools and healing scores taken from the serial photographs.

DETAILED DESCRIPTION:
This is a randomised controlled pilot study to assess the feasibility of copper impregnated stockings. All patients with CEAP classification 4 in both legs and venous disease identified by venous duplex will be recruited from the vascular clinics within Croydon Health Services over a period of three months. All patients will be given a patient information sheet describing the study prior to consent. Patients will be giving adequate time to read the information. Informed consent and the agreement for photography of their legs will be obtained. Patients will be assessed at baseline and at 2, 4 and 8 weeks follow-up.

Copper impregnated stockings:

All patients will be asked to wear compression stockings (14-18mmHg). These closed-toe and below-the-knee stockings are made of 88% nylon, 5% elastin, and 7% spandex and come in various sizes. One of the pair will have copper oxide ions permanently attached to the nylon fibres and these stockings will contain 2-3% copper ions. The patients will wear a copper stocking on one leg (study leg) and a non-copper stocking on the other (control leg). Both the patients and the clinicians will be blinded to the copper impregnated stocking.

Randomisation:

All stockings are marked with an 'L' for the left or 'R' for the right foot. The manufacturer has randomly marked the copper stockings with an 'L' or 'R' and paired these with a non-copper stocking. A closed envelope will contain the unique numbers of all the pairs of stockings and the information on which sock contains the copper. This envelope will remain closed for the whole recruitment period.

Patient data, history and physical examination:

Demographic data such as age, ethnicity, height and weight will be collected. Past medical history such as concomitant (chronic) diseases and the use of medications will be obtained. At each visit, subjective symptoms will be obtained using the Aberdeen Varicose Veins Questionnaire (AVVQ). For obtaining objective signs, the CEAP classification and the Venous Clinical Severity Scoring (VCSS) will be performed for grading the severity of the venous insufficiency per leg individually, and photographs with the Eykona® 3D camera will be taken. All data sets will be coded and anonymised. The data will be stored in a secure room within the Trust. All electronic data will be stored within password protected IT system within the Trust, which is only accessible by the clinical and research team.

Eykona® Wound Measurement System:

Skin changes associated with lipodermatosclerosis such as erythema, induration, hyperpigmentation and white atrophy, will be measured using the Eykona® Wound Measuring System (Type EYK10001). This system contains a 3D portable camera with software that enables precise measurements of wound size and tissue condition. Photographs will be taken at each visit. The surface area of the skin changes will be calculated.

Statistical analysis:

Statistical analysis will be performed using SPSS version 20.0 or higher. The CEAP classification, the Venous Clinical Severity Score and the AVVQ score at the 2, 4, and 8 weeks assessment will be compared with the baseline scores. The length, width and surface area of the skin condition from the leg with the copper will be compared with the control leg and the measurements at the 2, 4, and 8 weeks assessment will be compared with the baseline measurements. Paired t-test will be used for continuous data at baseline and a multilevel (mixed) regression model will be used to analyse the change over time.

Sample size calculation:

The sample size for this study will be 15. This number is based on the prevalence of the disease in this hospital over three months' time. There is no existing data available to allow a sample size calculation. The data collection of this pilot study will enable power calculation for a larger multicentre study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* CEAP classification 4 in both legs
* Venous disease confirmed by venous duplex
* Ability to understand and read the patient information sheet (in English)
* Ability to give informed consent

Exclusion Criteria:

* Inability to give consent
* Pregnancy
* Current ulceration
* Wilson's disease
* Allergy to copper
* Arterial insufficiency of the lower extremities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Aberdeen Varicose Vein Questionnaire (AVVQ) | 2 weeks
  Validated questionnaire consisting of 13 questions on signs and symptoms of chronic venous insufficiency for each leg seperately and questions on compression stocking usage and quality of life. The scoring of the questionnaire is from 0, which indicates no effect on the patient, to 100, which indicates a severe effect.
Venous Clinical Severity Scoring (VCSS) | 24 hours
  Assessment tool consisting of 10 items: pain, varicose veins, oedema, skin pigmentation, inflammation, induration, ulceration (number, size and duration) and use of compression therapy, which are scored on a severity scale from 0 to 3.

SECONDARY OUTCOMES:
Lipodermatosclerosis surface area | 2, 4 and 8 weeks after wearing compression stockings
  Surface area of the affected skin measured using 3D photographs with the Eykona® Wound Measuring System (Type EYK10001).

CONTACTS AND LOCATIONS:
Overall Officials: Abdul H Sultan, Principal Investigator — Croydon Health Services NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rabe E, Guex JJ, Puskas A, Scuderi A, Fernandez Quesada F; VCP Coordinators. Epidemiology of chronic venous disorders in geographically diverse populations: results from the Vein Consult Program. Int Angiol. 2012 Apr;31(2):105-15. PMID 22466974
- [Background] Van den Oever R, Hepp B, Debbaut B, Simon I. Socio-economic impact of chronic venous insufficiency. An underestimated public health problem. Int Angiol. 1998 Sep;17(3):161-7. PMID 9821029
- [Background] Motykie GD, Caprini JA, Arcelus JI, Reyna JJ, Overom E, Mokhtee D. Evaluation of therapeutic compression stockings in the treatment of chronic venous insufficiency. Dermatol Surg. 1999 Feb;25(2):116-20. doi: 10.1046/j.1524-4725.1999.08095.x. PMID 10037516
- [Background] Eklof B, Perrin M, Delis KT, Rutherford RB, Gloviczki P; American Venous Forum; European Venous Forum; International Union of Phlebology; American College of Phlebology; International Union of Angiology. Updated terminology of chronic venous disorders: the VEIN-TERM transatlantic interdisciplinary consensus document. J Vasc Surg. 2009 Feb;49(2):498-501. doi: 10.1016/j.jvs.2008.09.014. PMID 19216970
- [Background] Raju S, Hollis K, Neglen P. Use of compression stockings in chronic venous disease: patient compliance and efficacy. Ann Vasc Surg. 2007 Nov;21(6):790-5. doi: 10.1016/j.avsg.2007.07.014. PMID 17980798
- [Background] Borkow G, Gabbay J. Copper as a biocidal tool. Curr Med Chem. 2005;12(18):2163-75. doi: 10.2174/0929867054637617. PMID 16101497
- [Background] O'Gorman J, Humphreys H. Application of copper to prevent and control infection. Where are we now? J Hosp Infect. 2012 Aug;81(4):217-23. doi: 10.1016/j.jhin.2012.05.009. Epub 2012 Jun 26. PMID 22738611
- [Background] Borkow G, Gabbay J, Zatcoff RC. Could chronic wounds not heal due to too low local copper levels? Med Hypotheses. 2008;70(3):610-3. doi: 10.1016/j.mehy.2007.06.006. Epub 2007 Aug 6. PMID 17689198
- [Background] Sen CK, Khanna S, Venojarvi M, Trikha P, Ellison EC, Hunt TK, Roy S. Copper-induced vascular endothelial growth factor expression and wound healing. Am J Physiol Heart Circ Physiol. 2002 May;282(5):H1821-7. doi: 10.1152/ajpheart.01015.2001. PMID 11959648
- [Background] Tenaud I, Sainte-Marie I, Jumbou O, Litoux P, Dreno B. In vitro modulation of keratinocyte wound healing integrins by zinc, copper and manganese. Br J Dermatol. 1999 Jan;140(1):26-34. doi: 10.1046/j.1365-2133.1999.02603.x. PMID 10215764
- [Background] Ahmed Z, Briden A, Hall S, Brown RA. Stabilisation of cables of fibronectin with micromolar concentrations of copper: in vitro cell substrate properties. Biomaterials. 2004 Feb;25(5):803-12. doi: 10.1016/s0142-9612(03)00596-9. PMID 14609669
- [Background] Uauy R, Olivares M, Gonzalez M. Essentiality of copper in humans. Am J Clin Nutr. 1998 May;67(5 Suppl):952S-959S. doi: 10.1093/ajcn/67.5.952S. PMID 9587135
- [Background] Hostynek JJ, Dreher F, Maibach HI. Human skin penetration of a copper tripeptide in vitro as a function of skin layer. Inflamm Res. 2011 Jan;60(1):79-86. doi: 10.1007/s00011-010-0238-9. Epub 2010 Aug 20. PMID 20721598
- [Background] Weinberg, I., Lazary, A., Jefidoff, A., Vatine, J.J., Borkow, G., Ohana, N. Safety of using diapers containing copper oxide in chronic care elderly patients. Open Biol J. 2013;6:54-59.
- [Background] Borkow G, Okon-Levy N, Gabbay J. Copper oxide impregnated wound dressing: biocidal and safety studies. Wounds. 2010 Dec;22(12):301-10. PMID 25901580
- [Derived] Arendsen LP, Vig S, Thakar R, Sultan AH. Impact of copper compression stockings on venous insufficiency and lipodermatosclerosis: A randomised controlled trial. Phlebology. 2019 May;34(4):224-230. doi: 10.1177/0268355518795329. Epub 2018 Aug 27. PMID 30149775

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03283800/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03283800/ICF_001.pdf